CLINICAL TRIAL: NCT03067688
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase3 Trial to Evaluate the Efficacy and Safety of Co-administrated Temisartan/Amlodipine and Rosuvastatin in Subjects With Hypertension and Hyperlipidemia
Brief Title: Clinical Trial of Temisartan/Amlodipine & Rosuvastatin in Subjects With Hypertension and Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YHP1604-301
Record Dates: First submitted 2017-02-01; First posted 2017-03-01 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Drug Combinations; telmisartan amlodipine combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Combination drug:Temisartan+Amlodipine+Rosuvastatin" (Experimental): 60 subjects will be assigned and the subjects will be administered "Temisartan+Amlodipine+Rosuvastatin" for 8 weeks.
  Interventions: Drug: Temisartan+Amlodipine+Rosuvastatin (Combination drug)
- Temisartan+Amlodipine (Active Comparator): 60 subjects will be assigned and the subjects will be administered "Twynsta Tab.(Temisartan+Amlodipine)" for 8 weeks.
  Interventions: Drug: Temisartan+Amlodipine
- Temisartan+Rosuvastatin (Active Comparator): 60 subjects will be assigned and the subjects will be administered "Micardis Tab. and Crestor Tab.(Temisartan+Rosuvastatin)" for 8 weeks.
  Interventions: Drug: Temisartan+Rosuvastatin

INTERVENTIONS:
Drug: Temisartan+Amlodipine+Rosuvastatin (Combination drug) — PO, Once daily(QD), 8weeks
  Other Names: Twynsta Tab.+Crestor Tab.
  Arms: "Combination drug:Temisartan+Amlodipine+Rosuvastatin"
Drug: Temisartan+Amlodipine — PO, Once daily(QD), 8weeks
  Other Names: Twynsta Tab.
  Arms: Temisartan+Amlodipine
Drug: Temisartan+Rosuvastatin — PO, Once daily(QD), 8weeks
  Other Names: Micardis Tab.+Crestor Tab.
  Arms: Temisartan+Rosuvastatin

SUMMARY:
Randomized, double-blind, active-controlled, multicenter phase 3 trial to evaluate efficacy and safety of co-administrated temisartan/amlodipine and rosuvastatin in subjects with hypertension and hyperlipidemia.

DETAILED DESCRIPTION:
This trial is a phase 3 study to evaluate efficacy and safety of co-administrated temisartan/amlodipine and rosuvastatin in subjects with hypertension and hyperlipidemia.

In "Temisartan/Amlodipine/Rosuvastatin" treatment group, 60 subjects will be assigned and the subjects administer "Temisartan/Amlodipine/Rosuvastatin" 8 for weeks.

In "Temisartan/Amlodipine" treatment group, 60 subjects will be assigned and the subjects administer "Temisartan/Amlodipine" for 8 weeks.

In "Temisartan/Rosuvastatin" treatment group, 60 subjects will be assigned and the subjects administer "Temisartan/Rosuvastatin" for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Subjects with hypertension and hyperlipidemia

Exclusion Criteria:

1. Patients with known or suspected secondary hypertension
2. Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Mean sitting systolic blood pressure (MSSBP) | Baseline, Week 8
  MSSBP change form the baseline at Week 8
Low density lipoprotein cholesterol (LDL-C) | Baseline, Week 8
  LDL-C change form the baseline at Week 8

SECONDARY OUTCOMES:
MSSBP (Mean sitting systolic blood pressure) | Baseline, Week 4
  MSSBP change form the baseline at Week 4
Mean sitting diastolic blood pressure (MSDBP) | Baseline, Week 4, Week 8
  MSDBP change form the baseline at Week 4, 8
Low density lipoprotein cholesterol (LDL-C) | Baseline, Week 4
  LDL-C change form the baseline at Week 4
Total Cholesterol (TC) | Baseline, Week 4, Week 8
  TC change form the baseline at Week 4, 8
High density lipoprotein cholesterol (HDL-C) | Baseline, Week 4, Week 8
  HDL-C change form the baseline at Week 4, 8
Low density lipoprotein cholesterol/High density lipoprotein cholesterol (LDL-C/HDL-C) | Baseline, Week 4, Week 8
  LDL-C/HDL-C change form the baseline at Week 4, 8
Total Cholesterol/High density lipoprotein cholesterol (TC/HDL-C) | Baseline, Week 4, Week 8
  TC/HDL-C change form the baseline at Week 4, 8
Triglyceride (TG) | Baseline, Week 4, Week 8
  TG change form the baseline at Week 4, 8

CONTACTS AND LOCATIONS:
Overall Officials: Hyunhee Na, MD, Study Director — Yuhan Corporation
Locations (1):
- Seoul Natuional University Hospital, Seoul, Jongno, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin X, Kim MH, Han KH, Hong SJ, Ahn JC, Sung JH, Cho JM, Lee HC, Choi SY, Lee K, Kim WS, Rhee MY, Kim JH, Hong SP, Yoo BS, Cho EJ, Lee JH, Kim PJ, Park CG, Hyon MS, Shin JH, Lee SH, Sung KC, Hwang J, Kwon K, Chae IH, Seo JS, Kim H, Lee H, Cho Y, Kim HS. Efficacy and safety of co-administered telmisartan/amlodipine and rosuvastatin in subjects with hypertension and dyslipidemia. J Clin Hypertens (Greenwich). 2020 Oct;22(10):1835-1845. doi: 10.1111/jch.13893. Epub 2020 Sep 16. PMID 32937023